CLINICAL TRIAL: NCT04380493
Title: Special Considerations for the Use of the Transient Elastography Paediatric Probe, Compared to the Standard M Probe, Indirect Serological Markers and Histology
Brief Title: The Use of the Transient Elastography Paediatric Probe, Compared to the M Probe, Indirect Biomarkers and Histology
Status: Completed | Type: Observational
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Jesús Quintero, Pediatric Hepatologist, physician, Hospital Vall d'Hebron
Other Study IDs: PR(AMI)147/2019
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Elastography; Fibrosis, Liver; Pediatrics; Chronic Liver Disease
Keywords: Elastography; liver biopsy; biopsy; indirect biomarkers
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: hepatic transient elastography using S probe and M probe
  Other Names: Compare results with liver biopsy; Calculate indirect fibrosis markers (APRI and FIB-4)

SUMMARY:
The purpose of this study is to assess the reliability, reproducibility and accuracy of the paediatric probe of transient elastography in detecting liver fibrosis in children, besides its limitations and side effects. At the same time, to assess whether indirect fibrosis markers are a valid tool to detect absence or mild fibrosis in paediatric patients

DETAILED DESCRIPTION:
A retrospective cohort study, including all patients younger than 18 years of age with chronic liver disease who underwent a transient elastography, was performed. The study was carried out in the joint Unit of Paediatric Complex Hepatology and Liver Transplant, encompassing two third level paediatric hospitals, between 2015 and 2019. The study protocol was approved by local ethic committee (identifier code: PR(AMI)147/2019) and informed consent was signed by patient's legal guardians and patients over 16 years old.

Liver stiffness was assessed with FibroScan® (Echosens, France, model 502, class IIa, year 2010), which was performed by an experienced operator to avoid interobserver bias and in the same standardized conditions (fasting, decubitus position, right arm in maximal abduction, transducer placed over the right lobe). S probe (model 8; 5 MHz; diameter 5 mm), that measures depths ranging from 15-50 mm (S1: 15-40 mm; S2: 20-50 mm), was selected if chest circumference (CC) < 75 cm (S1: ≤ 45 cm; S2: 45-75 cm). M probe (3.5 MHz; diameter 7 mm), measuring depths range 35-75mm, was used if CC ≥ 75 cm. Both probes met the calibration terms. Elastographic parameters studied were: stiffness (KPa), interquartile range (IQR) and success rate (SR). Adult-validated liver stiffness measurement ranges to classify the fibrosis degree were taken as a reference: F0-F1 (≤7.6 KPa), F2 (7.7-9.4 KPa), F3 (9.5-14 KPa) and F4 (>14 KPa). The examination was successful when the median of at least 10 valid values, had a SR higher than 60% and with an IQR/LSM lower than 30%.

The following sociodemographic, clinical and analytical data were collected: age, sex, underlying liver disease and analytical parameters (alanine aminotransferase (ALT) U/L, aspartate aminotransferase (AST) U/L, gamma glutamyl transferase (GGT) U/L, total bilirubin (mg/dl), cholesterol (mg/dl), platelets (109/L), prothrombin time (%)). The following liver fibrosis test Scores were calculated using the obtained data:

* Fibrosis 4 Score (FIB-4) = Age (years) x AST (U/L) / platelets (109/L) x √ALT (U/L).
* AST to Platelet Radio Index (APRI) = AST (upper normal limit) (UI/l)/ platelets x 109 x 100.

Eighteen clinically indicated liver biopsies were performed and staged according METAVIR score (F0-F4). Blood test, fibrosis scores and biopsies were performed within 6 months of transient elastography. No clinical or analytical changes were observed during this period.

The Faces Pain Scale was used for assessing pain severity. Statistical analysis: Kolmogorov-Smirnov test checked out if variables followed a normal distribution. Continuous variables are presented as mean ± standard deviation or median (interquartile range) and categorical variables as number of subjects and percentage. Correlation between continuous variables were calculated using Pearson's and Spearman's correlation coefficient. The variance's analysis (ANOVA) and the Kruskal Wallis test were used to compare qualitative with quantitative variables. Two-tailed p-Values of <0.05 were considered as statistically significant. Sensitivity, specificity, positive predictive value and negative predictive value were calculated in the assessment of FIB-4 and APRI as a diagnostic test to detect absence or mild fibrosis (F0-F1), using the results obtained by TE as a reference. The statistical analyses were performed with SPSS software (v. 21, SPSS Inc., Chicago, IL, USA) and Prism (v. 7.04 GraphPad Software Inc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 18 years of age with chronic liver disease who underwent a transient elastography.
* Parents / legal guardians and the patients themselves, if applicable, have read, understood and signed the informed consent of the study.

Exclusion Criteria:

* Patients who do not meet all the inclusion criteria for inclusion in the study protocol.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients of both sexes, aged 0 months to 18 years, suffering from various chronic liver diseases.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Validation of FibroScan's® pediatric (S) probe in children | 4 years
  To describe our experience with FibroScan's® pediatric (S) probe; its reliability, reproducibility, and accuracy in detecting fibrosis, as compared to M probe and histology, as well as its limitations and side effects

SECONDARY OUTCOMES:
Validation of indirect fibrosis markers | 4 years
  To assess whether indirect fibrosis markers (APRI and FIB-4) are a valid tool to detect absence or mild fibrosis in paediatric patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roulot D, Czernichow S, Le Clesiau H, Costes JL, Vergnaud AC, Beaugrand M. Liver stiffness values in apparently healthy subjects: influence of gender and metabolic syndrome. J Hepatol. 2008 Apr;48(4):606-13. doi: 10.1016/j.jhep.2007.11.020. Epub 2008 Jan 3. PMID 18222014
- [Background] Friedrich-Rust M, Ong MF, Martens S, Sarrazin C, Bojunga J, Zeuzem S, Herrmann E. Performance of transient elastography for the staging of liver fibrosis: a meta-analysis. Gastroenterology. 2008 Apr;134(4):960-74. doi: 10.1053/j.gastro.2008.01.034. Epub 2008 Jan 18. PMID 18395077
- [Background] Bamber J, Cosgrove D, Dietrich CF, Fromageau J, Bojunga J, Calliada F, Cantisani V, Correas JM, D'Onofrio M, Drakonaki EE, Fink M, Friedrich-Rust M, Gilja OH, Havre RF, Jenssen C, Klauser AS, Ohlinger R, Saftoiu A, Schaefer F, Sporea I, Piscaglia F. EFSUMB guidelines and recommendations on the clinical use of ultrasound elastography. Part 1: Basic principles and technology. Ultraschall Med. 2013 Apr;34(2):169-84. doi: 10.1055/s-0033-1335205. Epub 2013 Apr 4. PMID 23558397
- [Background] Cosgrove D, Piscaglia F, Bamber J, Bojunga J, Correas JM, Gilja OH, Klauser AS, Sporea I, Calliada F, Cantisani V, D'Onofrio M, Drakonaki EE, Fink M, Friedrich-Rust M, Fromageau J, Havre RF, Jenssen C, Ohlinger R, Saftoiu A, Schaefer F, Dietrich CF; EFSUMB. EFSUMB guidelines and recommendations on the clinical use of ultrasound elastography. Part 2: Clinical applications. Ultraschall Med. 2013 Jun;34(3):238-53. doi: 10.1055/s-0033-1335375. Epub 2013 Apr 19. PMID 23605169
- [Background] Sterling RK, Lissen E, Clumeck N, Sola R, Correa MC, Montaner J, S Sulkowski M, Torriani FJ, Dieterich DT, Thomas DL, Messinger D, Nelson M; APRICOT Clinical Investigators. Development of a simple noninvasive index to predict significant fibrosis in patients with HIV/HCV coinfection. Hepatology. 2006 Jun;43(6):1317-25. doi: 10.1002/hep.21178. PMID 16729309
- [Background] Wai CT, Greenson JK, Fontana RJ, Kalbfleisch JD, Marrero JA, Conjeevaram HS, Lok AS. A simple noninvasive index can predict both significant fibrosis and cirrhosis in patients with chronic hepatitis C. Hepatology. 2003 Aug;38(2):518-26. doi: 10.1053/jhep.2003.50346. PMID 12883497
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140
- [Background] Fitzpatrick E, Quaglia A, Vimalesvaran S, Basso MS, Dhawan A. Transient elastography is a useful noninvasive tool for the evaluation of fibrosis in paediatric chronic liver disease. J Pediatr Gastroenterol Nutr. 2013 Jan;56(1):72-6. doi: 10.1097/MPG.0b013e31826f2760. PMID 22922372
- [Background] de Ledinghen V, Le Bail B, Rebouissoux L, Fournier C, Foucher J, Miette V, Castera L, Sandrin L, Merrouche W, Lavrand F, Lamireau T. Liver stiffness measurement in children using FibroScan: feasibility study and comparison with Fibrotest, aspartate transaminase to platelets ratio index, and liver biopsy. J Pediatr Gastroenterol Nutr. 2007 Oct;45(4):443-50. doi: 10.1097/MPG.0b013e31812e56ff. PMID 18030211
- [Background] Tokuhara D, Cho Y, Shintaku H. Transient Elastography-Based Liver Stiffness Age-Dependently Increases in Children. PLoS One. 2016 Nov 18;11(11):e0166683. doi: 10.1371/journal.pone.0166683. eCollection 2016. PMID 27861607
- [Background] Cho Y, Tokuhara D, Morikawa H, Kuwae Y, Hayashi E, Hirose M, Hamazaki T, Tanaka A, Kawamura T, Kawada N, Shintaku H. Transient Elastography-Based Liver Profiles in a Hospital-Based Pediatric Population in Japan. PLoS One. 2015 Sep 23;10(9):e0137239. doi: 10.1371/journal.pone.0137239. eCollection 2015. PMID 26398109
- [Background] Menten R, Leonard A, Clapuyt P, Vincke P, Nicolae AC, Lebecque P. Transient elastography in patients with cystic fibrosis. Pediatr Radiol. 2010 Jul;40(7):1231-5. doi: 10.1007/s00247-009-1531-z. Epub 2010 Feb 5. PMID 20135110
- [Background] Engelmann G, Gebhardt C, Wenning D, Wuhl E, Hoffmann GF, Selmi B, Grulich-Henn J, Schenk JP, Teufel U. Feasibility study and control values of transient elastography in healthy children. Eur J Pediatr. 2012 Feb;171(2):353-60. doi: 10.1007/s00431-011-1558-7. Epub 2011 Aug 23. PMID 21861093
- [Background] Goldschmidt I, Streckenbach C, Dingemann C, Pfister ED, di Nanni A, Zapf A, Baumann U. Application and limitations of transient liver elastography in children. J Pediatr Gastroenterol Nutr. 2013 Jul;57(1):109-13. doi: 10.1097/MPG.0b013e31829206a0. PMID 23539048
- [Background] Alkhouri N, Sedki E, Alisi A, Lopez R, Pinzani M, Feldstein AE, Nobili V. Combined paediatric NAFLD fibrosis index and transient elastography to predict clinically significant fibrosis in children with fatty liver disease. Liver Int. 2013 Jan;33(1):79-85. doi: 10.1111/liv.12024. Epub 2012 Nov 12. PMID 23146095
- [Background] Lee CK, Perez-Atayde AR, Mitchell PD, Raza R, Afdhal NH, Jonas MM. Serum biomarkers and transient elastography as predictors of advanced liver fibrosis in a United States cohort: the Boston children's hospital experience. J Pediatr. 2013 Oct;163(4):1058-64.e2. doi: 10.1016/j.jpeds.2013.04.044. Epub 2013 Jun 5. PMID 23759423
- [Background] Fung J, Lee CK, Chan M, Seto WK, Wong DK, Lai CL, Yuen MF. Defining normal liver stiffness range in a normal healthy Chinese population without liver disease. PLoS One. 2013 Dec 26;8(12):e85067. doi: 10.1371/journal.pone.0085067. eCollection 2013. PMID 24386446
- [Background] Nobili V, Vizzutti F, Arena U, Abraldes JG, Marra F, Pietrobattista A, Fruhwirth R, Marcellini M, Pinzani M. Accuracy and reproducibility of transient elastography for the diagnosis of fibrosis in pediatric nonalcoholic steatohepatitis. Hepatology. 2008 Aug;48(2):442-8. doi: 10.1002/hep.22376. PMID 18563842
- [Background] Rubio A, Monpoux F, Huguon E, Truchi R, Triolo V, Rosenthal-Allieri MA, Deville A, Rosenthal E, Boutte P, Tran A. Noninvasive procedures to evaluate liver involvement in HIV-1 vertically infected children. J Pediatr Gastroenterol Nutr. 2009 Nov;49(5):599-606. doi: 10.1097/MPG.0b013e3181a15b72. PMID 19668009
- [Background] Vinciguerra T, Brunati A, David E, Longo F, Pinon M, Ricceri F, Castellino L, Piga A, Giraudo MT, Tandoi F, Cisaro F, Dell Olio D, Isolato G, Romagnoli R, Salizzoni M, Calvo PL. Transient elastography for non-invasive evaluation of post-transplant liver graft fibrosis in children. Pediatr Transplant. 2018 Mar;22(2). doi: 10.1111/petr.13125. Epub 2018 Jan 25. PMID 29369488
- [Background] Lee CK, Mitchell PD, Raza R, Harney S, Wiggins SM, Jonas MM. Validation of Transient Elastography Cut Points to Assess Advanced Liver Fibrosis in Children and Young Adults: The Boston Children's Hospital Experience. J Pediatr. 2018 Jul;198:84-89.e2. doi: 10.1016/j.jpeds.2018.02.062. PMID 29685617
- [Background] Kim S, Kang Y, Lee MJ, Kim MJ, Han SJ, Koh H. Points to be considered when applying FibroScan S probe in children with biliary atresia. J Pediatr Gastroenterol Nutr. 2014 Nov;59(5):624-8. doi: 10.1097/MPG.0000000000000489. PMID 25003372
- [Background] Shen QL, Chen YJ, Wang ZM, Zhang TC, Pang WB, Shu J, Peng CH. Assessment of liver fibrosis by Fibroscan as compared to liver biopsy in biliary atresia. World J Gastroenterol. 2015 Jun 14;21(22):6931-6. doi: 10.3748/wjg.v21.i22.6931. PMID 26078570
- [Background] Goldschmidt I, Stieghorst H, Munteanu M, Poynard T, Schlue J, Streckenbach C, Baumann U. The use of transient elastography and non-invasive serum markers of fibrosis in pediatric liver transplant recipients. Pediatr Transplant. 2013 Sep;17(6):525-34. doi: 10.1111/petr.12116. Epub 2013 Jun 27. PMID 23802661
- [Background] Myers RP, Pomier-Layrargues G, Kirsch R, Pollett A, Duarte-Rojo A, Wong D, Beaton M, Levstik M, Crotty P, Elkashab M. Feasibility and diagnostic performance of the FibroScan XL probe for liver stiffness measurement in overweight and obese patients. Hepatology. 2012 Jan;55(1):199-208. doi: 10.1002/hep.24624. Epub 2011 Nov 18. PMID 21898479
- [Background] de Ledinghen V, Vergniol J, Foucher J, El-Hajbi F, Merrouche W, Rigalleau V. Feasibility of liver transient elastography with FibroScan using a new probe for obese patients. Liver Int. 2010 Aug;30(7):1043-8. doi: 10.1111/j.1478-3231.2010.02258.x. Epub 2010 May 14. PMID 20492500
- [Background] Friedrich-Rust M, Hadji-Hosseini H, Kriener S, Herrmann E, Sircar I, Kau A, Zeuzem S, Bojunga J. Transient elastography with a new probe for obese patients for non-invasive staging of non-alcoholic steatohepatitis. Eur Radiol. 2010 Oct;20(10):2390-6. doi: 10.1007/s00330-010-1820-9. Epub 2010 Jun 6. PMID 20526777
- [Background] Kim SY, Seok JY, Han SJ, Koh H. Assessment of liver fibrosis and cirrhosis by aspartate aminotransferase-to-platelet ratio index in children with biliary atresia. J Pediatr Gastroenterol Nutr. 2010 Aug;51(2):198-202. doi: 10.1097/MPG.0b013e3181da1d98. PMID 20531020
- [Background] McGoogan KE, Smith PB, Choi SS, Berman W, Jhaveri R. Performance of the AST-to-platelet ratio index as a noninvasive marker of fibrosis in pediatric patients with chronic viral hepatitis. J Pediatr Gastroenterol Nutr. 2010 Mar;50(3):344-6. doi: 10.1097/MPG.0b013e3181aed725. PMID 20118806
- [Background] Leung DH, Khan M, Minard CG, Guffey D, Ramm LE, Clouston AD, Miller G, Lewindon PJ, Shepherd RW, Ramm GA. Aspartate aminotransferase to platelet ratio and fibrosis-4 as biomarkers in biopsy-validated pediatric cystic fibrosis liver disease. Hepatology. 2015 Nov;62(5):1576-83. doi: 10.1002/hep.28016. Epub 2015 Sep 28. PMID 26223427
- [Background] Yang HR, Kim HR, Kim MJ, Ko JS, Seo JK. Noninvasive parameters and hepatic fibrosis scores in children with nonalcoholic fatty liver disease. World J Gastroenterol. 2012 Apr 7;18(13):1525-30. doi: 10.3748/wjg.v18.i13.1525. PMID 22509085
- [Background] Mansoor S, Yerian L, Kohli R, Xanthakos S, Angulo P, Ling S, Lopez R, Christine CK, Feldstein AE, Alkhouri N. The evaluation of hepatic fibrosis scores in children with nonalcoholic fatty liver disease. Dig Dis Sci. 2015 May;60(5):1440-7. doi: 10.1007/s10620-014-3494-7. Epub 2014 Dec 25. PMID 25540086
- [Background] Andersen SB, Ewertsen C, Carlsen JF, Henriksen BM, Nielsen MB. Ultrasound Elastography Is Useful for Evaluation of Liver Fibrosis in Children-A Systematic Review. J Pediatr Gastroenterol Nutr. 2016 Oct;63(4):389-99. doi: 10.1097/MPG.0000000000001171. PMID 26925609